CLINICAL TRIAL: NCT03522792
Title: The Effect of Neurotensin on Appetite, Food Intake, Blood Glucose Regulation, Hormone Secretion, and the Degradation of Neurotensin in Vivo
Brief Title: Neurotensin - an Important Regulator of Appetite in Humans?
Acronym: NIRAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Simon Veedfald, Principal investigator, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: Neurotensin BMI/HH 2017 UCPH
Record Dates: First submitted 2017-12-14; First posted 2018-05-11 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Physiology - Regulation of Appetite and Food Intake
Keywords: food intake; appetite; obesity treatment; neurotensin; gastrointestinal; peptide
MeSH Terms: interventions — Neurotensin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be studied on multiple occasions (5 days) in a randomised and double blinded fashion. One day will serve as an acclimatization day.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will not be informed of the nature of the infusion they are administered on any of the study days. The investigator will be provided with an infusion (either isotonic saline with HSA or isotonic salin with HSA + neurotensin) prepared by a designated colleague
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Saline + ad libitum meal (Experimental): This will serve as the placebo / control day for the NT + ad libitum meal study day.
  Interventions: Other: Saline; Other: Ad libitum meal
- NT + ad libitum meal (Experimental): Neurotensin (NT) infusion followed by an ad libitum meal to study the effect of NT on ad libitum food intake.
  Interventions: Other: Neurotensin; Other: Ad libitum meal
- Saline + liquid meal + ad libitum meal (Experimental): Saline infusion followed a standardized liquid mixed meal followed by an ad libitum meal. This will serve as the placebo / control day for the NT + standardized liquid mixed meal + ad libitum meal study day. Investigating the effect of NT on the second meal effect.
  Interventions: Other: Saline; Other: Ad libitum meal; Other: Liquid meal
- NT + liquid meal + ad libitum meal (Experimental): NT infusion followed a standardized liquid mixed meal followed by an ad libitum meal. This study day aims to study the effect of NT on the second meal effect.
  Interventions: Other: Neurotensin; Other: Ad libitum meal; Other: Liquid meal
- Neurotensin (Experimental): Acclimatization day
  Interventions: Other: Neurotensin; Other: Ad libitum meal

INTERVENTIONS:
Other: Neurotensin — Intravenous infusion of neurotensin
  Arms: NT + ad libitum meal; NT + liquid meal + ad libitum meal; Neurotensin
Other: Saline — Intravenous infusion of saline
  Arms: Saline + ad libitum meal; Saline + liquid meal + ad libitum meal
Other: Ad libitum meal — Participants will be served a large meal serving. They will be instructed to eat until they do not feel hungry anymore.
Other: Liquid meal — A standardized mixed liquid meal will be ingested to stimulate endogenous peptide hormone release
  Arms: NT + liquid meal + ad libitum meal; Saline + liquid meal + ad libitum meal

SUMMARY:
Neurotensin (NT) is a gut peptide released postprandially from the small intestine. It is known to exert a range of enterogastrone effects and in animal models it reduces food intake when administered by parenteral routes.

This study investigates whether the anorexic effects of NT suggested by animal studies can be translated.

ELIGIBILITY:
Inclusion Criteria:

* age = or above 18 years
* normal haemoglobin levels
* male
* informed consent

Exclusion Criteria:

* Diabetes mellitus (fasting plasma glucose or HbA1c)
* Familiy history of diabetes mellitus
* Intestinal disease (incl e.g. inflammatory bowel disease and malabsorbtion)
* Family history of inflammatory bowel disease
* Previous intestinal resection
* Body mass index (BMI) over 25 kg/m2
* Smoker
* Nephropathy (S-creatinine> 130 μM)
* Liver disease (ALAT and/or ASAT > 2 × upper normal limit)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Ad libitum food intake (ad libitum days) | 60 min
  Neurotensin (NT) and saline will be infused on two occasions in random order, double blinded. After 1h of infusion an ad libitum meal will be served. When the meal is completed food intake will be determined by weighing the leftovers.
Ad libitum food intake (liquid meal + ad libitum days) | 240 min
  Neurotensin (NT) and saline will be infused on two occasions in random order, double blinded. 1h into the infusions a standardized liquid mixed meal will be ingested. After another 180 min an ad libitum meal will be served. When the meal is completed food intake will be determined by weighing the leftovers.

SECONDARY OUTCOMES:
Appetite and gastrointestinal sensations (ad libitum days) | -60, -15, 15, 30, 60, 90, 120 min
  Using visual analogue scales (VAS) the effect of infusions and meals will be documented.
  Ad libitum meals will also be evaluated using VAS.
Appetite and gastrointestinal sensations (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Using visual analogue scales (VAS) the effect of infusions and meals will be documented.
  Ad libitum meals will also be evaluated using VAS.
Plasma glucose (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Bed-side measurements of plasma glucose
Plasma glucose (liquid meal + ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 180, 240 min
  Bed-side measurements of plasma glucose
Neurotensin (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Plasma analysis
Neurotensin (liquid meal + ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 180, 240 min
  Plasma analysis
Insulin (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Serum analysis
Bile acids (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Plasma analysis
bile acids (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis
Ghrelin (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Plasma analysis
Ghrelin (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis
Glucagon-like peptide-1 (GLP-1) (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Plasma analysis
Glucagon-like peptide-1 (GLP-1) (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis
Glucose-dependent insulinotropic polypeptide (GIP) (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis
Peptide YY (PYY) (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis
Paracetamol (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Serum analyses
Pancreatic polypeptide (PP) (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis
Pancreatic polypeptide (PP) (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Plasma analysis
Cholecystokinin (CCK) (ad libitum days) | -60, -30, -15, -1, 0- , 15, 30, 45, 60, 75, 90, 105, 120 min
  Plasma analysis
Cholecystokinin (CCK) (liquid meal + ad libitum days) | -60, -15, 15, 60, 90, 120, 150, 180, 210, 240 min
  Plasma analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Capital, Denmark

IPD SHARING:
Plan to Share IPD: No